CLINICAL TRIAL: NCT06662786
Title: A Randomized, Open-label Phase 3 Study of Amivantamab and mFOLFOX6 or FOLFIRI Versus Cetuximab and mFOLFOX6 or FOLFIRI as First-line Treatment in Participants With KRAS/NRAS and BRAF Wild-type Unresectable or Metastatic Left-sided Colorectal Cancer
Brief Title: A Study of Amivantamab and mFOLFOX6 or FOLFIRI Versus Cetuximab and mFOLFOX6 or FOLFIRI as First-line Treatment in Participants With KRAS/NRAS and BRAF Wild-type Unresectable or Metastatic Left-sided Colorectal Cancer
Acronym: OrigAMI-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372COR3001; 61186372COR3001 (Other: Janssen Research & Development, LLC); 2024-513852-13-00 (Registry Identifier: EUCT number)
Expanded Access: NCT04599712 (Approved for marketing)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — amivantamab; Cetuximab; Fluorouracil; Leucovorin; Levoleucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Amivantamab in Combination With Chemotherapy (Experimental): Participants will receive amivantamab in combination with chemotherapy (mFOLFOX6 [chemotherapy consisting of 5-fluorouracil, leucovorin calcium (folinic acid) or levoleucovorin, and oxaliplatin] or FOLFIRI [chemotherapy consisting of 5-fluorouracil, leucovorin calcium (folinic acid) or levoleucovorin, and irinotecan hydrochloride]) for 28-days treatment cycles and will continue to receive the treatment until radiographic disease progression or other discontinuation criteria are met.
  Interventions: Biological: Amivantamab; Drug: 5-fluorouracil; Drug: Leucovorin calcium/Levoleucovorin; Drug: Oxaliplatin; Drug: Irinotecan Hydrochloride
- Arm B: Cetuximab in Combination With Chemotherapy (Active Comparator): Participants will receive cetuximab in combination with chemotherapy (mFOLFOX6 or FOLFIRI) for 28-days treatment cycles and will continue to receive the treatment until radiographic disease progression or other discontinuation criteria are met.
  Interventions: Biological: Cetuximab; Drug: 5-fluorouracil; Drug: Leucovorin calcium/Levoleucovorin; Drug: Oxaliplatin; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Biological: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372
  Arms: Arm A: Amivantamab in Combination With Chemotherapy
Biological: Cetuximab — Cetuximab will be administered.
  Other Names: Erbitux
  Arms: Arm B: Cetuximab in Combination With Chemotherapy
Drug: 5-fluorouracil — 5-fluorouracil will be administered as chemotherapy regimen.
Drug: Leucovorin calcium/Levoleucovorin — Leucovorin calcium/Levoleucovorin will be administered as chemotherapy regimen.
Drug: Oxaliplatin — Oxaliplatin will be administered as chemotherapy regimen.
Drug: Irinotecan Hydrochloride — Irinotecan hydrochloride will be administered as chemotherapy regimen.

SUMMARY:
The purpose of this study is to compare how long the participants are disease-free (progression-free survival) when treated with amivantamab and chemotherapy with 5-fluorouracil, leucovorin calcium (folinic acid) or levoleucovorin, oxaliplatin (mFOLFOX6) or 5-fluorouracil, leucovorin calcium (folinic acid) or levoleucovorin, and irinotecan hydrochloride (FOLFIRI) versus cetuximab and mFOLFOX6 or FOLFIRI in adult participants with Kirsten rat sarcoma viral oncogene homolog (KRAS)/ Neuroblastoma RAS viral oncogene homolog (NRAS) and v-Raf murine sarcoma viral oncogene homolog B1 (BRAF) wild type (WT) unresectable or metastatic left-sided colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed adenocarcinoma of the left-sided colorectal cancer. Participants must have unresectable or metastatic disease
* Determined to have Kirsten rat sarcoma viral oncogene (KRAS), neuroblastoma RAS viral oncogene homolog (NRAS), and v-raf murine sarcoma viral oncogene homolog B (BRAF) wild-type (WT) tumor by local and/or central testing (if available)
* Must agree to the submission of fresh tumor tissue
* Have measurable disease according to RECIST v1.1
* Have an eastern cooperative oncology group (ECOG) performance status (PS) of 0 or 1

Exclusion Criteria:

* Has medical history of (noninfectious) interstitial lung disease (ILD) /pneumonitis/pulmonary fibrosis or has current ILD/pneumonitis/pulmonary fibrosis, or where suspected ILD/pneumonitis/pulmonary fibrosis cannot be ruled out by imaging at screening
* Has known allergies, hypersensitivity, or intolerance to excipients of any of the following: (a) amivantamab or cetuximab, (b) any component of mFOLFOX6 and, (c) any component of FOLFIRI
* Has a prior or concurrent second malignancy other than the disease under study or one whose natural history or treatment is likely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Participant with known mismatch repair deficiency (dMMR)/ high microsatellite instability (MSI-H) status and human epidermal growth factor receptor 2 (HER2)-positive/amplified tumor
* Has prior exposure to any agents that target epidermal growth factor receptor (EGFR) or mesenchymal epithelial transition (MET)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) | Up to 4 years and 2 months
  PFS is defined as the time from randomization until the date of objective disease progression or death (due to any cause), whichever comes first, as assessed by BICR using response evaluation criteria in solid tumors (RECIST) version (v) 1.1. Participants who have not progressed or have not died at the time of analysis will be censored at their last evaluable RECIST v1.1 assessment date.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 7 Years 3 Months
  OS is defined as the time from the date of randomization to the date of participant's death due to any cause. Any participant not known to have died at the time of analysis will be censored based on the last recorded date on which the participant was known to be alive.
Objective Response Rate (ORR) as Assessed by BICR | Up to 7 Years 3 Months
  ORR is defined as the percentage of randomized participants achieving complete response (CR) or partial response (PR), as determined by BICR using RECIST v1.1 criteria. On or before the date of subsequent systemic anticancer therapy or date of curative-intent procedure, whichever occurs first.
Progression Free Survival (PFS) as Assessed by Investigator | Up to 7 Years 3 Months
  PFS is defined as the time from randomization until the date of objective disease progression or death (due to any cause), whichever comes first, as assessed by the investigator. Participants who have not progressed or have not died at the time of analysis will be censored at their last evaluable disease assessment date.
Objective Response Rate (ORR) as Assessed by Investigator | Up to 7 Years 3 Months
  ORR is defined as the percentage of randomized participants achieving complete CR or PR, as assessed by the investigator.
Duration of Response (DOR) as Assessed by BICR | Up to 7 Years 3 Months
  DOR is defined as time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR, as assessed by BICR using RECIST v1.1 criteria.
Duration of Response (DOR) as Assessed Investigator | Up to 7 Years 3 Months
  DOR is defined as time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR, as assessed by the investigator.
Progression-free Survival After Subsequent Therapy (PFS2) | Up to 7 Years 3 Months
  PFS2 is defined as the time from randomization until the date of second objective disease progression, after initiation of subsequent anticancer therapy, based on investigator assessment (after that used for PFS) or death, whichever comes first.
Disease Control Rate (DCR) as Assessed by BICR | Up to 7 Years 3 Months
  DCR is defined as the percentage of randomized participants achieving CR, PR, or stable disease (with minimum duration of 7 weeks) as assessed by BICR using RECIST v1.1 criteria.
Disease Control Rate (DCR) as Assessed by Investigator | Up to 7 Years 3 Months
  DCR is defined as the percentage of randomized participants achieving CR, PR, or stable disease (with minimum duration of 7 weeks) as assessed by the investigator.
Time to Treatment Failure | Up to 7 Years 3 Months
  Time to treatment failure is defined as time from randomization to discontinuation of therapy for any reason including death, progression, toxicity, or initiation of new anticancer therapy.
Curative Resection (R0) Rate | Up to 7 Years 3 Months
  Curative resection (R0) rate is defined as the percentage of the full analysis set who underwent curative-intent surgery a where the residual tumor classification was R0.
Number of Participants with Adverse Events (AEs) by Severity | Up to 7 Years 3 Months
  An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. AE severity will be graded according to the national cancer institute common terminology criteria for adverse events (NCI-CTCAE) v5.0. by using the standard grades as follows: Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; and Grade 5: Death related to AE.
Number of Participants with Abnormalities in Laboratory Values | Up to 7 Years 3 Months
  Participants with abnormalities in laboratory values (such as serum chemistry, hematology) will be reported.
Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | From Baseline up to 7 Years 3 Months
  The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the health-related quality of life (HRQoL) of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status / quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Time to Worsening in Symptoms and Functioning as Measured by EORTC QLQ-C30 | Up to 7 Years 3 Months
  The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status / quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptom.
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer Module 29 (EORTC-QLQ-C30) Score | From Baseline up to 7 Years 3 Months
  The EORTC QLQ-CR29, is a self-administered, 29-item questionnaire measuring the HRQoL of participants with colorectal cancer. The QLQ CR29 includes items that evaluate symptoms (gastrointestinal, urinary, pain, and others) and functional areas (sexual, body image, weight, and anxiety) that are associated with colorectal cancer and its treatments. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". All scores are linearly converted into a scale from 0 to 100. Higher scores indicate greater functioning and more severe symptoms.
Time to Worsening in Symptoms and Functioning as Measured by EORTC QLQ-CR29 | Up to 7 Years 3 Months
  The EORTC QLQ-CR29, is a self-administered, 29-item questionnaire measuring the HRQoL of participants with colorectal cancer. The QLQ CR29 includes items that evaluate symptoms (gastrointestinal, urinary, pain, and others) and functional areas (sexual, body image, weight, and anxiety) that are associated with colorectal cancer and its treatments. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". All scores are linearly converted into a scale from 0 to 100. Higher scores indicate greater functioning and more severe symptoms.
Overall Side Effect Burden as Measured by European Organisation for Research and Treatment of Cancer (EORTC) Item 168 Scale Score | Up to 7 Years 3 Months
  The EORTC item 168 is a single item used to measure the overall impact of treatment side effects. Responses are rated on a 4-point Likert response scale ranging from 1 "not at all" to 4 "very much." Higher scores indicate severe side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (228):
- United States (70):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - CBCC Global Research, Bakersfield, California
  - Los Angeles Cancer Network, Glendale, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Torrance Memorial Physicians Network, Torrance, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown Univ Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists South, Fort Myers, Florida
  - AdventHealth Medical Group Oncology and Hematology at Orlando, Orlando, Florida
  - Florida Cancer Specialists North Region, St. Petersburg, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Illinois CancerCare, Peoria, Illinois
  - Fort Wayne Medical Oncology & Hematology, Fort Wayne, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Start Midwest, Grand Rapids, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists Midwest Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Astera Cancer Care, East Brunswick, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Perlmutter Cancer Center at NYU Long Island, Mineola, New York
  - Mount Sinai, New York, New York
  - Mount Sinai West, New York, New York
  - NYU Langone Medical Center NYU Hematology Associates, New York, New York
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center Fairview Hospital Moll Pavilion, Cleveland, Ohio
  - Taussig Cancer Insititute Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic Cancer Center Independence Family Health Center, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Hillcrest Hospital, Mayfield Heights, Ohio
  - Cleveland Clinic Cancer Centers Sandusky, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Cleveland Clinic Cancer Center South Pointe Hospital, Warrensville Heights, Ohio
  - Wooster Milltown Specialty and Surgery Center, Wooster, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology West Texas, Abilene, Texas
  - Texas Oncology DFW, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Baylor Scott and White Health, Temple, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
  - Inova Schar Cancer Institute Dept of Fairfax Hospital, Fairfax, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute, Edmonds, Washington
  - Swedish Cancer Institute, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - William S. Middleton Memorial VA, Madison, Wisconsin
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - Hopital de Jolimont, Haine Saint Paul La Louviere
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Brazil (11):
  - Fundacao Pio XII, Barretos
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Hospital Santa Izabel Santa Casa de Misericordia da Bahia, Salvador
  - Clinica de Hematologia e Oncologia Viver Ltda, Santa Maria
  - Fundacao Faculdade Regional De Medicina S Jose Rio Preto Hospital De Base, São José do Rio Preto
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Associacao Feminina de Educacao e Combate ao Cancer Hospital Santa Rita de Cassia, Vitória
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
- China (22):
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Hunan Cancer hospital, Changsha
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The Sixth Affiliated Hospital Sun Yat sen University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Central People's Hospital, Huizhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - West China Hospital of Sichuan University, Sichuan
  - First Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
- France (9):
  - Institut Sainte Catherine, Avignon
  - Hopital Claude Huriez, Lille
  - Hopital Prive Jean Mermoz, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hopital Saint Antoine, Paris
  - Hopital Haut Leveque, Pessac
  - CHU De Poitiers, Poitiers
  - Gustave Roussy, Villejuif
- Germany (10):
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Essen University Hospital, Essen
  - Krankenhaus NorthWest, Frankfurt am Main
  - Praxis fur interdisziplinare Onkologie & Hamatologie GbR, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - National Center for Tumor Diseases NCT, Heidelberg
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Klinikum der Universitaet Muenchen, Munich
  - Universitatsklinikum Ulm, Ulm
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem, Szeged
- India (5):
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi
  - B P Poddar Hospital and Medical research Limited, Kolkata
  - Tata Memorial Hospital, Mumbai
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre, Varanasi
- Israel (7):
  - Yitzhak Shamir Medical Center, Beer Yaakov
  - Rambam Medical Center, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta MC, Tel Aviv
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Dei Tumori Di Milano, Milan
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
- Japan (9):
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - Aichi Cancer Center, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - The University of Osaka Hospital, Suita
  - The Cancer Institute Hospital of JFCR, Tokyo
- Malaysia (7):
  - Hospital Canselor Tuanku Muhriz UKM, Cheras
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - National Cancer Institute, Putrajaya
- Netherlands (6):
  - Meander Medisch Centrum, Amersfoort
  - Antoni van Leeuwenhoek, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - UMC Utrecht, Utrecht
- Poland (9):
  - Bialostockie Centrum Onkologii im Marii Sklodowskiej Curie w Bialymstoku, Bialystok
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut BadawczyOddz w Gliwicach, Gliwice
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - SPZOZ Ministerstwa Spraw Wewnetrznych z Warminsko Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - SPZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarowskiego, Opole
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Pan American Center for Oncology Trials LLC, Barrio Monacillos, Puerto Rico
- South Korea (6):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (8):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skanes universitetssjukhus, Lund
  - Sodersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala University, Uppsala
- Taiwan (5):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Bakirkoy Training and Research Hospital, Istanbul
  - Marmara University Pendik Training Hospital, Istanbul
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Sakarya University Training and Research Hospital, Sakarya
- United Kingdom (9):
  - Birmingham Heartlands Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Castle Hill Hospital, Hull
  - St James University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Mount Vernon Cancer Centre, Northwood
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency